CLINICAL TRIAL: NCT07370922
Title: Glucagon-Like Peptide 1 Receptor Agonist in Diabetes Mellitus Management in Children and Adolescents With Transfusion-Dependent Thalassemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran yousef, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MS 794/2024
Record Dates: First submitted 2026-01-09; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Transfusion Dependent Beta Thalassemia
Keywords: GLP-1 receptor agonist; Dulaglutide; Diabetes; Transfusion Dependent Thalassemia
MeSH Terms: conditions — Diabetes Mellitus | interventions — dulaglutide; Control Groups; Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dulaglutide group (Experimental)
  Interventions: Drug: Dulaglutide 0.75Mg/0.5Ml Inj Pen
- Control group (Active Comparator): Control group
  Interventions: Drug: control group (insulin)

INTERVENTIONS:
Drug: Dulaglutide 0.75Mg/0.5Ml Inj Pen — Dulaglutide subcutaneous injection in a dose of 0.75 mg once weekly for 6 months.
  Arms: Dulaglutide group
Drug: control group (insulin) — Insulin basal blocs according to guidelines
  Arms: Control group

SUMMARY:
Blood transfusion and iron-chelation therapy have prolonged and improved the quality of life in patients with β-thalassemia. The improvement was mainly due to the decrease in mortality from heart failure Such a treatment, however, leads to chronic iron overload and frequently to endocrine complications, especially the development of diabetes.

The prevalence of diabetes mellitus (DM) in β-thalassemia varies from 9.7% to 29% and the overall prevalence of impaired fasting glucose (IFG) and impaired glucose tolerance (IGT) is 17.2% and 12.4% respectively in transfusion dependent thalassemia (TDT) patients.

GLP-1 is a proglucagon derived peptide that is released from gut endocrine cells in response to nutrient intake. This molecule is rapidly inactivated by the action of dipeptidyl peptidase IV (DPP-4) which limits its use as therapeutic agent.

Recent guidelines by the American Diabetes Association and the European Association for the Study of Diabetes recommend that for patients with type 2 diabetes, GLP-1 receptor agonists (GLP-1RAs) are preferable to insulin as the initial injection therapy and are also the preferred choice for addition to basal insulin for combination injection therapy.

An increasing number of clinical trials of agents in youth-onset T2D resulted in the availability of more efficacy data and regulatory approval for two Glucagon-like peptide-1 (GLP-1) receptor agonists (Liraglutide and Exenatide) in Pediatrics.

The Efficacy of the daily GLP-1 agonist, Liraglutide, in youth-onset T2D wasstudied in the Ellipse trial, which demonstrated placebo-subtracted. HbA1c lowering of 1% and 1.5% at 26 and 52 weeks, respectively. This glycemic reduction was accompanied by a small decrease in BMI z-score. Liraglutide (Victoza 0.6-1.8 mg a day) subsequently received approval by the FDA for use in youth 12-17 years of age.

Recently, extended release exenatide (Bydureon BCise 2 mg) was approved as a once-weekly injection for youth 10-17 years of age based on data from the BCB114 study showing superiority to placebo in lowering HbA1c with a between-group difference of 0.85 percentage points.

Hence, the aim of this study is to assess the efficacy and safety of GLP-1 receptor agonist versus conventional insulin therapy in the management of diabetes mellitus in children with transfusion -dependent Thalassemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-18 years old.
2. Children with TDT according to the Thalassemia International Federation (TIF) guidelines (Farmakis et al., 2022).
3. Children with diabetes mellitus according to the International Society for Pediatric and Adolescent Diabetes (ISPAD) 2022 guidelines (Libman et al., 2022).

Exclusion Criteria:

1. Other hemoglobinopathies as alpha thalassemia or sickle thalassemia patients.
2. Other disorders that may affect glucose homeostasis rather than β-TM.
3. Autoimmune disease, collagen diseases, hypo- or hyper-thyroidism, infections, tumors, hematological diseases other than β-TM.
4. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN 2).
5. Intake of any vitamins or food supplements one month before study and participation in a previous investigational drug study within the three months preceding screening.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Change in glycemic variability using continuous glucose monitoring after 6 months. | 6 months
  Change in glycemic variability using continuous glucose monitoring after 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No